CLINICAL TRIAL: NCT04635761
Title: The Roswell AIR (Awareness, Information and Resources for Lung Cancer Screening) Program: A Community-Partnered Lung Cancer Screening Intervention
Brief Title: Awareness, Information, and Resources for Lung Cancer Screening Program for Community-Partnered Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 781020; NCI-2020-08297 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 781020 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-11-05; First posted 2020-11-19 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (AIR Program) (Experimental): Participants complete the Roswell Awareness, Information and Resources for Lung Cancer Screening (AIR) Program over 45 minutes and then receive the High-Risk Lung Cancer Tip Sheet..
  Interventions: Behavioral: Educational Intervention; Behavioral: Questionnaire Administration

INTERVENTIONS:
Behavioral: Educational Intervention — Complete AIR Program and receive the High-Risk Lung Cancer Tip Sheet
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Behavioral: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial investigates an educational program called Awareness, Information, and Resources for Lung Cancer Screening Program in improving knowledge about lung cancer screening in medically underserved communities. This program aims to educate and remove barriers to lung cancer screening among medically underserved community members who are eligible for lung cancer screening, and to improve access to evidence-based screening guidelines for early detection for lung cancer in the Western New York area.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Collaborate with community organizations and leaders to leverage community-based assets to disseminate education about lung cancer screening.

II. Reach medically underserved, high risk community members. III. Enhance lung cancer screening knowledge among medically underserved, high risk community members.

IV. Navigate screening-eligible community members to lung cancer screening.

OUTLINE:

Participants complete the Roswell Awareness, Information and Resources for Lung Cancer Screening (AIR) Program over 45 minutes and then receive the High-Risk Lung Cancer Tip Sheet.

ELIGIBILITY:
Inclusion Criteria:

* Members of all races and ethnic groups are eligible for this study

Exclusion Criteria:

* Adults unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Number of programs offered | Up to 1 year
Average number of attendees at each site | Up to 1 year
Demographics of attendees at each site | Up to 1 year
Number of medically underserved, high risk community members reached | Up to 1 year
Percent change in lung cancer screening awareness as assessed before and after program completion | Up to 1 year
  Pre and post questionnaire to be given to participants
Percent change in knowledge of eligibility guidelines for screening as assessed before and after program completion | Up to 1 year
  Pre and post questionnaire to be given to participants before and after educational sessions
Percent Change in knowledge of benefits of early detection as assessed before and after program completion | Up to 1 year
  Pre and post questionnaire to be completed by participants before and after educational sessions
Change in fear, worry, and increased health-related self-efficacy | Up to 1 year
  Pre and post questionnaire to be completed by participants before and after educational sessions
Number of screening eligible individuals reached | Up to 1 year
Number of screening eligible individuals navigated to lung cancer screening | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bouchard, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States